CLINICAL TRIAL: NCT01815190
Title: Retrospective Analysis of Frequency of Systemic Involvement in IgA-positive Cutaneous Immune Complex Vasculitis Versus IgA-negative Cutaneous Immune Complex Vasculitis
Brief Title: IgA-positive Versus IgA-negative Immune Complex Vasculitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Muenster (Other)
Responsible Party: Principal Investigator, Cord Sunderkötter, Professor Dr, University Hospital Muenster
Other Study IDs: 2011-040-f-S
Record Dates: First submitted 2013-03-18; First posted 2013-03-20 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Cutaneous Vasculitis
Keywords: immune complex vasculitis; cutaneous vasculitis; IgA vasculitis; IgA nephropathy
MeSH Terms: conditions — Skin Diseases, Vascular; IgA Vasculitis; Glomerulonephritis, IGA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- IgA-positive vasculitis: Patients with immune complex vasculitis who show perivascular deposits of IgA
- IgA-negative vasculitis: Patients with immune complex vasculitis who show no perivascular deposits of IgA

SUMMARY:
Cutaneous vasculitis due to vascular deposition of large circulating immune complexes is a disease frequently seen by general practitioners and dermatologists. The clinical symptom is palpable purpura with predilection for the lower legs.

In some cases vasculitis also affects systemic organs, such as the kidneys and the intestine.

When the immune complexes contain immunoglobulin class A (IgA) and when there is systemic involvement, the disease has been referred to as Henoch Schönlein purpura.

When there are no signs of systemic involvement, the disease has been referred to as cutaneous leukocytoclastic angiitis.

The investigators hypothesize that palpable purpura with predilection for lower legs is a pathognomonic clinical sign for immune complex vasculitis in both IgA vasculitis and IgA-negative vasculitis, but that only the presence of IgA in immune complexes is likely to be associated with systemic involvement and therefore warrants more extensive diagnostic procedures Vice versa the investigators postulate that the presence of IgG or IgM without IgA in immune complexes excludes systemic involvement The investigators also want to investigate to which of the 2 groups patients with palpable purpura and negative immunofluorescence should be assigned.

ELIGIBILITY:
Inclusion Criteria:

* histologically proven leukocytoclastic vasculitis
* clinically palpable purpura

Exclusion Criteria:

* no histological confirmation
* relevant data missing in file

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients of the department of dermatology in Muenster with histologically proven leukocytoclastic vasculitis in files in last 10-20 years
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2011-01; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Frequency of systemic involvement in patients with IgA-positive versus patients with non-IgA-positive immune complex vasculitis | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Cord Sunderkoetter, Prof Dr MD, Principal Investigator — Department of Dermatology, Univ Hospital of Muenster
Locations (1):
- Department of Dermatology, Univ hospital of Muenster, Münster, Germany